CLINICAL TRIAL: NCT03046563
Title: The Effectiveness of the Applying of Acupressure and Abdominal Massage to Improving Constipation in Stroke Patients.
Brief Title: The Applying of Acupressure and Abdominal Massage to Improving Constipation in Stroke Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Li-Li Chen (Other)
Responsible Party: Sponsor-Investigator, Li-Li Chen, China Medical University, China Medical University Hospital
Organization: China Medical University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MOST 105-2314-B-039-033 -
Record Dates: First submitted 2017-02-05; First posted 2017-02-08 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Acupressure; Abdominal Massage; Constipation; Stroke Patients
Keywords: acupressure; abdominal massage; constipation; stroke patients; Traditional Chinese medicine
MeSH Terms: conditions — Constipation | interventions — Acupressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupressure and Abdominal Massage (Experimental): Pressing the Hegu (LI 4), Zusanli (ST 36) , Tianshu(ST 25) and abdominal massage for eight minutes total, press once in the morning and afternoon, seven days total and two days for follow the trail.
  Interventions: Other: Acupressure and Abdominal Massage
- Pressing the sham points (Sham Comparator): Pressing the sham points for eight minutes total, press once in the morning and afternoon, seven days total and two days for follow the trail.
  Interventions: Other: Pressing the Sham points

INTERVENTIONS:
Other: Acupressure and Abdominal Massage — Pressing the Hegu (LI 4), Zusanli (ST 36) , Tianshu(ST 25) and abdominal massage for eight minutes
  Arms: Acupressure and Abdominal Massage
Other: Pressing the Sham points — Pressing the sham points for eight minutes
  Other Names: the Sham points
  Arms: Pressing the sham points

SUMMARY:
Experimental research design with two-group repeated-measure design. Experimental group was pressing the Hegu (LI 4), Zusanli (ST 36) , Tianshu(ST 25) and abdominal massage for eight minutes total, press once in the morning and afternoon, seven days total and two days for follow the trail. Control group was pressing sham ponits. Research tools to self semi-structured questionnaire collected data on patient's diet, activity, medication, defecation patterns, subjective defecation feelingauscultation bowel sounds like.

DETAILED DESCRIPTION:
Experimental research design with two-group repeated-measure design. The investigators estimate there are recruit fifty patients from related rehabilitation hospital of a medical center in Taichung, central Taiwan, using randomization put patients in experimental group and control group. Experimental group Pressing the Hegu (LI 4), Zusanli (ST 36) , Tianshu(ST 25) and abdominal massage for eight minutes total, press once in the morning and afternoon, seven days total and two days for follow the trail. Control group was pressing sham ponits. Research tools to self semi-structured questionnaire collected data on patient's diet, activity, medication, defecation patterns, subjective defecation feelings, and auscultation bowel sounds like. The investigators expected the results of this study can provide clinical nursing care for stroke patients of reference, to improve quality of care, and increase acupressure to improve the empirical data of stroke in patients with constipation.

ELIGIBILITY:
Inclusion Criteria:

1. patients who were diagnosed as stroke, and in stability phase.
2. patients who had constipation symptoms.
3. patients whose platelets counts more than 150,000 / μ.

Exclusion Criteria:

1. Consciousness is not clear.
2. The physician diagnosed with irritable bowel syndrome.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
defecation patterns | 9 days
  measure defecation frequency and nature

SECONDARY OUTCOMES:
auscultation bowel sounds | 9 days
  auscultation bowel sounds before and after intervention

IPD SHARING:
Plan to Share IPD: No